CLINICAL TRIAL: NCT01385722
Title: Molecular Analysis of Thoracic Malignancies
Status: Enrolling by invitation | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-21319; SU-06232011-7986 (Other: Stanford University); THOR0004 (Other: OnCore)
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Thymus Cancer; Thymoma; Thymic Carcinoma; Lung Cancer; Carcinoma, Non-Small-Cell Lung; Mesothelioma
MeSH Terms: conditions — Thymus Neoplasms; Thymoma; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Mesothelioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The potential tumor tissues to be collected include paraffin-embedded tissue, frozen tissues, or fresh tissue. These will be stored in conjunction with the Stanford Tissue Bank.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A research study to learn about the biologic features of cancer development, growth, and spread. We are studying components of blood, tumor tissue, normal tissue, and other fluids, such as urine, cerebrospinal fluid, abdominal or chest fluid in patients with cancer. Our analyses of blood, tissue, and/or fluids may lead to improved diagnosis and treatment of cancer by the identification of markers that predict clinical outcome, markers that predict response to specific therapies, and the identification of targets for new therapies.

DETAILED DESCRIPTION:
In the United States, an estimated 222,520 lung and bronchus cancers will be diagnosed in 2010, and 157,300 people will die of this disease. Therefore, there is an urgent need for safer and more effective therapies for lung cancer.1 Lung cancer falls into two major classifications, non-small cell lung cancer (NSCLC) which accounts for approximately 87%, and small cell lung cancer (SCLC), which accounts for the remainder. Thymomas are the most common tumors of the anterior mediastinum, and typically occur in adults older than 40 years. While surgical resection and radiation often effectively treat these tumors, a minority continue to progress and eventually lead to death. Thymic carcinomas are a related subset of tumors that more often metastasize and are more aggressive. Finally, mesothelioma often behaves as aggressively as lung cancer, and is not frequently amenable to curative resection.

While the role of molecular alterations has yet to be defined in the treatment of SCLC, thymoma, and mesothelioma, there is an increasing recognition that molecular alterations in NSCLC are important predictors of response to novel targeted therapies. Small molecule tyrosine kinase inhibitors (TKI) of the epidermal growth factor receptor (EGFR) signaling pathway, such as erlotinib and gefitinib, improve survival in the second-line treatment of unselected patients with NSCLC. However, retrospective subgroup analysis of these clinical trials has revealed that patients with particular clinical features were more likely to benefit from therapy, such as those with tumors of adenocarcinoma histology, women, Asian ethnicity, and light or never smokers. Conventional Deoxyribonucleic acid (DNA) sequencing of tumors from multiple series of patients that had dramatic responses to gefitinib, as compared with patients without responses, revealed the presence of characteristic genetic mutations in the EGFR gene.4-6 The previously identified clinical markers of response to EGFR TKIs were found to be commonly associated with the presence of these mutations; thus, these clinical features are actually believed to be surrogates for the molecular biomarker of EGFR mutation. Over 90% of EGFR tyrosine kinase domain mutations associated with sensitivity to EGFR Tyrosine kinase inhibitor (TKI) therapy fall into two categories, in-frame deletions in exon 19, and the L858R point mutation in exon 21. These mutations appear to specifically activate both cell proliferation, via activation of the MAP kinase pathway, and survival signals, via activation of the PI3 kinase pathway.7 Therefore, tumors with EGFR mutations are "oncogene addicted" to EGFR survival signals, relying exclusively upon the EGFR signaling cascade to maintain viability, which explains their exquisite sensitivity to TKI therapy. A number of recent large randomized studies have conclusively demonstrated that clinical selection of patients alone is inadequate, and instead establish EGFR mutation status as the single most important predictive marker of response to EGFR-TKI therapy.8-10 In another emerging but similar story, genetic fusion of the anaplastic lymphoma kinase (ALK) tyrosine kinase to a partner protein, EML4, appears to strongly predict sensitivity to the ALK TKI, crizotinib. 11 In addition, there is evidence that less common mutations in NSCLC, such as BRAF mutations and ERBB2 (e.g. HER2) mutations, may also predict response to targeted therapies.

In summary, identification of genetic alterations in NSCLC is increasingly essential for individualizing treatments and performing molecular diagnostics. While the investigators do not anticipate benefits to individual patients, identification of molecular alterations in small cell lung cancer, thymic malignancies, and mesothelioma may provide similar keys to the utilization of novel therapies. This project aims to create a registry of patients and tumors to further the characterization of molecular alterations in thoracic malignancies and develop markers of early detection.

ELIGIBILITY:
Inclusion Criteria:

1.Histologically proven diagnosis of non-small cell lung cancer, small cell lung cancer, thymoma, thymic carcinoma, mesothelioma, or carcinoma of unknown primary consistent with the presentation of a primary thoracic malignancy.

2.18 years of age or older.

3.Ability to understand and the willingness to sign a written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified who come to the Stanford Cancer Center seeking a Thoracic Oncology medical opinion for their disease.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-08; Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Collect detailed clinical information on patients with thoracic malignancies via the electronic medical record and a detailed patient questionnaire | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neal, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States